CLINICAL TRIAL: NCT00036023
Title: A Randomized, Open-Label, Dose-Timing Study of Darbepoetin Alfa Administered Once Every 3 Weeks (Q3W) by Subcutaneous (SC) Injection for Treatment of Anemia in Subjects With Non-Myeloid Malignancies Receiving Multicycle Chemotherapy
Brief Title: Chemotherapy Related Anemia in Patients With Non-Myeloid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20010162; NCT00039247 (obsolete NCT alias)
Record Dates: First submitted 2002-05-07; First posted 2002-05-08 (Estimated); Last update posted 2009-05-11 (Estimated); Status verified 2009-05

CONDITIONS: Lymphoma; Breast Neoplasms; Lung Neoplasms; Multiple Myeloma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma; Breast Neoplasms; Lung Neoplasms; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa

SUMMARY:
Chemotherapy can often cause anemia in patients with cancer. Anemia is a low number of red blood cells. The symptoms of anemia may include fatigue, dizziness, headache, chest pain, and shortness of breath. Erythropoietin is a hormone made by the kidneys that signals the bone marrow to produce more red blood cells. Recombinant human erythropoietin has been produced in the laboratory and has the same effect as the hormone produced by the body. Use of recombinant human erythropoietin allows the body to produce more red blood cells, possibly eliminating or decreasing your symptoms and the need for a red blood cell transfusion. Recombinant human erythropoietin is FDA approved to treat anemia in cancer patients receiving chemotherapy. This clinical study is investigating the effectiveness of darbepoetin alfa for the treatment of anemia in patients with non-myeloid malignancies who are receiving chemotherapy every three weeks. Darbepoetin alfa is a recombinant erythropoietic protein that stimulates the production of red blood cells. This medication has not been approved to treat cancer patients with anemia, however it has been approved by the FDA to treat chronic renal failure patients with anemia.

ELIGIBILITY:
* Patients with non-myeloid malignancies * Patients receiving at least 12 weeks of chemotherapy on a 3-week cycle schedule * Patients with anemia (hgb >/= 9.0 and </= 11.0 g/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Glaspy J, Henry D, Patel R, Tchekmedyian S, Applebaum S, Berdeaux D, Lloyd R, Berg R, Austin M, Rossi G; Darbepoetin Alfa 20010162 Study Group. Effects of chemotherapy on endogenous erythropoietin levels and the pharmacokinetics and erythropoietic response of darbepoetin alfa: a randomised clinical trial of synchronous versus asynchronous dosing of darbepoetin alfa. Eur J Cancer. 2005 May;41(8):1140-9. doi: 10.1016/j.ejca.2005.01.021. Epub 2005 Apr 8. PMID 15911237
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20010162.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/